CLINICAL TRIAL: NCT07310134
Title: An Open-Label, Multicenter Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Dose Escalation and Dose Expansion of ZX-8177 Tablets in Chinese Patients With Advanced Solid Tumors
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of ZX-8177 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX-8177-201; CTR20254582 (Other: http://www.chinadrugtrials.org.cn)
Record Dates: First submitted 2025-12-02; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Dose Escalation Phase:
  The specific design is as follows: starting dose is 100 mg BID, with a total of 5 predefined dose groups (100 mg BID, 200 mg BID, 400 mg BID, 800 mg BID, and 1200 mg BID).
  Interventions: Drug: ZX-8177

INTERVENTIONS:
Drug: ZX-8177 — Dose Escalation Phase:
  The starting dose is 100 mg BID, with a total of 5 predefined dose groups (100 mg BID, 200 mg BID, 400 mg BID, 800 mg BID, and 1200 mg BID).

SUMMARY:
This study is an open-label, multicenter, phase I clinical trial involving dose escalation and dose expansion of ZX-8177 in patients with advanced unresectable, recurrent, or metastatic solid tumors.

The study consists of two stages: dose escalation and dose expansion. It primarily aims to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), biomarkers, and preliminary efficacy of ZX-8177 as a monotherapy with continuous administration in Chinese patients with advanced solid tumors who have failed standard treatment or lack standard treatment options. The study also seeks to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD)/optimal biological dose (OBD), or recommended phase II dose (RP2D).

DETAILED DESCRIPTION:
Dose Escalation Phase:

The specific design is as follows:

The starting dose is 100 mg BID, with a total of five predefined dose groups (100 mg BID, 200 mg BID, 400 mg BID, 800 mg BID, and 1200 mg BID).

The trial employs an accelerated titration combined with a "3+3" dose escalation design:

For the first two dose groups (100 mg BID and 200 mg BID), one subject each will initially be enrolled for accelerated titration and dose escalation. If the enrolled subject in either group does not experience a Grade 2 or higher non-disease-related toxicity event (excluding asymptomatic laboratory abnormalities judged by the investigator to require no intervention) from the first dose administration until the end of the first cycle (the DLT observation period), the trial for the next dose group will proceed. If a DLT occurs, the escalation method will switch to the "3+3" dose escalation approach.

Starting from the 400 mg BID dose group, three subjects will initially be enrolled in each dose group. If no DLT is observed in the three subjects of a given dose group during the DLT observation period, the clinical trial for the next predefined escalated dose group will proceed.

If one of the three subjects in a dose group experiences a DLT during the DLT observation period, an additional three subjects will be enrolled in that dose group. If no DLT is observed among the newly enrolled three subjects, three subjects may be enrolled for the next higher dose group. If one or more DLTs are observed among the newly enrolled three subjects, that dose group is defined as the DLT dose group. No additional subjects may be enrolled in this group, and the dose escalation phase will conclude. The previous dose will then be determined as the Maximum Tolerated Dose (MTD). Enrollment in the DLT dose group must not exceed six subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in this clinical trial, understand and comply with the study procedures, and voluntarily sign the Informed Consent Form (ICF).
* 2. No gender restriction, age ≥ 18 years at the time of signing ICF.
* 3. Minimum expected survival period ≥ 3 months (as determined by the investigator's assessment).
* 4. ECOG score is 0-1.
* 5. Advanced malignant tumors confirmed by histology/cytology: Advanced solid tumors without standard effective treatment options, or those that are ineffective or recurrent after standard treatment, or intolerant to standard treatment, or for which standard treatment is not applicable at this stage.
* 6. The subject must have at least one measurable lesion defined by RECIST v1.1, which has not been previously irradiated or has shown clear disease progression after radiotherapy.
* 7.Adequate Organ Function:

  1. Renal: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min [Cockcroft-Gault formula: ([140 - age] × weight [kg] × [0.85 for females only]) / (72 × creatinine (mg/dl))]; qualitative urine protein ≤ 1+; if qualitative urine protein ≥ 2+, a 24-hour urine protein quantification test is required, and a result of <1 g is acceptable.
  2. Hepatic: AST and ALT ≤ 2.5 × ULN (for subjects with liver involvement, AST and ALT ≤ 4 × ULN); total bilirubin ≤ 1.5 × ULN (for subjects with Gilbert's syndrome, total bilirubin ≤ 3 × ULN). Coagulation function: For subjects not receiving anticoagulant therapy, the International Normalized Ratio (INR) and activated partial thromboplastin time (APTT) should be ≤ 1.5 × ULN.
  3. Bone Marrow: Absolute neutrophil count (ANC) > 1.5 × 10⁹/L; hemoglobin level ≥ 90 g/L; platelet count ≥ 90 × 10⁹/L (administration of medications with leukocyte/platelet-boosting effects within 14 days prior to enrollment to meet eligibility criteria is not permitted).
* 8. Female patients of childbearing potential must have a negative serum pregnancy test during screening. Female patients not of childbearing potential (meeting at least one of the following criteria):

  1. Have undergone hysterectomy or bilateral oophorectomy/salpingectomy, or
  2. Have medically confirmed ovarian failure, or
  3. Are medically confirmed to be physiologically postmenopausal (with amenorrhea for at least 12 consecutive months, excluding causes such as chemotherapy, radiotherapy, or the use of estrogen/progestin therapy or other pathological factors).
* 9. Females of childbearing potential and male partners of females of childbearing potential must agree to use effective contraception during the study and for 6 months (for females) or 3 months (for males) after the last dose of ZX-8177:

  1. Including prescription hormonal oral contraceptives, contraceptive injections, contraceptive patches, vaginal rings, intrauterine devices, barrier methods (e.g., condoms, diaphragms, or cervical caps), or spermicidal foams, creams, or gels, or
  2. Practice complete abstinence, or
  3. The sole sexual partner of a female of childbearing potential is a male who has been confirmed sterile.
* 10. Males must agree to avoid sperm donation during the study and for 3 months after the last dose of ZX-8177.

Exclusion Criteria:

* 1. Previous use of ENPP1 inhibitors or STING agonists.
* 2. Received anti-tumor drug treatment within 28 days prior to the first administration of the study drug (including small-molecule targeted drugs, oral fluorouracil-based chemotherapy drugs, or modern traditional Chinese medicine preparations approved by the National Medical Products Administration (NMPA) for anti-tumor therapy within 14 days; mitomycin C or nitrosourea-based chemotherapy drugs within 6 weeks), excluding bisphosphonates for bone metastases.
* 3. History of immune-related adverse events (irAEs) of grade ≥3 during previous immunotherapy.
* 4. Undergone radiotherapy within 14 days prior to the first administration of the study drug; palliative radiotherapy for the purpose of alleviating local symptoms (non-target lesion irradiation or local administration to non-target lesions) completed within one week before study enrollment is allowed.
* 5. Participation in any other interventional clinical trials within 1 month prior to enrollment or within less than 5 half-lives (except for subjects who have completed other clinical studies and are only undergoing subsequent survival follow-up).
* 6. History of any organ transplantation, including allogeneic stem cell transplantation, except for transplants that do not require immunosuppression (e.g., corneal transplantation, hair transplantation).
* 7. Major surgery requiring general anesthesia, liver ablation, or hepatic arterial intervention within 28 days before the first administration of the investigational drug; or surgery requiring local/epidural anesthesia within 2 weeks prior to starting the investigational drug; or the subject has planned surgery or is considered by the investigator to require surgery; or unresolved postoperative complications before dosing (major surgery is defined as procedures under general anesthesia or involving significant incisions);
* 8. Adverse reactions from prior anti-tumor therapy or complications/sequelae from surgery > Grade 1 or not resolved to baseline (CTCAE v5.0, except alopecia or other toxicities deemed by the investigator to pose no safety risk to the subject);
* 9. Administration of live, inactivated, or attenuated vaccines within 30 days before the first dose of the investigational drug; examples of live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, COVID, bacillus Calmette-Guérin (BCG), and typhoid vaccines; inactivated or attenuated vaccines such as injectable seasonal influenza vaccines, intranasal influenza vaccines (e.g., FluMist®), etc.;
* 10. Subjects with symptomatic central nervous system metastases or carcinomatous meningitis (including leptomeningeal carcinomatosis); if CNS metastases are present, they must be assessed by the investigator as asymptomatic and stable for at least 3 months.
* 11. History of another malignancy within the past 5 years, except malignancies treated with surgery alone and in continuous disease-free survival; except early-stage in situ carcinoma after resection;
* 12. Uncontrolled electrolyte disturbances (e.g., hypocalcemia, hypomagnesemia, hypokalemia);
* 13. Dysphagia;
* 14. Clinically uncontrolled pleural effusion, pericardial effusion, or ascites;
* 15. Systemic use of immunosuppressive doses (prednisone >10 mg/day or equivalent) of medications (e.g., corticosteroids) within 2 weeks before starting the investigational drug, excluding topical glucocorticoids via nasal spray, inhalation, or other local routes, or physiological doses of systemic glucocorticoids (i.e., not exceeding 10 mg/day prednisone or equivalent of other glucocorticoids);
* 16. Clinically significant active cardiac disease or history, including but not limited to any of the following:

  1. History of long QT syndrome or confirmed family history of long QT syndrome;
  2. History of clinically significant ventricular arrhythmias;
  3. History of unstable angina, acute myocardial infarction, coronary artery bypass grafting, or symptomatic congestive heart failure within 6 months before enrollment;
  4. Current implantable defibrillator or pacemaker for ventricular arrhythmias;
  5. Known concomitant medications required that prolong the QT interval;
  6. Baseline QTcF interval corrected by Fridericia's formula >450 msec (male) or >470 msec (female);
  7. Complete left bundle branch block or complete right bundle branch block with left anterior fascicular block (bifascicular block);
  8. Left ventricular ejection fraction (LVEF) <50% on echocardiography;
  9. Myocardial infarction, bypass, stent surgery, or other cardiac conditions deemed unsuitable for enrollment by the investigator within 6 months before dosing;
* 17. Underlying diseases that may interfere with study evaluation, such as:

  1. Poorly controlled hypertension (defined as resting systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥95 mmHg despite treatment with two or more antihypertensive agents of different mechanisms);
  2. Baseline hemoglobin A1c >8.0%;
* 18. Active infection, including clinically uncontrolled active infectious diseases within 14 days before enrollment such as acute pneumonia, unexplained persistent fever, etc.; or meeting any of the following criteria: a) Positive human immunodeficiency virus (HIV) test or known history of acquired immunodeficiency syndrome; b) Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, defined as HBsAg positive with HBV DNA copies above the upper limit of normal, or HCV-Ab positive; c) Active tuberculosis (history of exposure or positive tuberculin test; accompanied by clinical and/or imaging manifestations); d) Positive treponemal antibody; e) Cytomegalovirus (CMV) infection, etc.

Note: Subjects with positive HBsAg and/or HBcAb who are stable after medication (HBV-DNA <500 IU/mL) and cured hepatitis C subjects (HCV-RNA PCR negative in patients with known HCV history within <6 months before starting ZX-8177) may be enrolled. Virological monitoring is required before dosing on Day 15 of Cycle 1 and before dosing on Day 1 of each subsequent cycle. Prophylactic antiviral therapy may be considered based on the subject's condition.

* 19. Known drug-induced liver injury, chronic active hepatitis, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cholangitis, persistent extrahepatic obstruction due to gallstones, cirrhosis, or portal hypertension;
* 20. Severe lung disease (history of or concurrent severe interstitial lung disease, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm);
* 21. Gastrointestinal dysfunction that may limit absorption of the investigational drug, including motility disorders, malabsorption syndromes, inflammatory bowel disease, chronic diarrhea, Crohn's disease, and/or prior surgery affecting absorption;
* 22. Psychiatric disorders or substance abuse;
* 23.Pregnant or breastfeeding women;
* 24. Allergic constitution or history of severe allergies;
* 25. Intolerance to venipuncture;
* 26. History of autoimmune disease, or active, known, or suspected autoimmune disorders (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune vasculitis, thyroid disorders, or glomerulonephritis). Subjects with the following conditions may be enrolled: vitiligo, type I diabetes, residual hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement, or conditions not expected to recur in the absence of external triggers;
* 27. Expected receipt of other systemic anti-tumor therapy during the study;
* 28. The patient is currently taking known inhibitors of OATP1B1, OATP1B3, and OAT3 and cannot discontinue use within 1 week before starting the investigational drug (or within 5 half-lives of the drug, whichever is longer) and during the study;
* 29. Any other condition considered by the investigator to be unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Participant Safety as characterized by frequency and severity of adverse events | Up to 30 days following last dose.
  Safety profile including frequency and severity of adverse events that are related to treatment.
In the dose escalation phase, the tolerability metric is to evaluate the incidence of dose related toxicity (DLT). | Up to 28 days following first dose.
  In the dose escalation phase, the tolerability metric is to evaluate the incidence of DLT.

SECONDARY OUTCOMES:
Changes in CCL4 during the treatment process | Up to 30 days following last dose.
  Changes in CCL4 during the treatment process
Objective Response Rate (ORR) | Up to 14 days following last dose.
  Defined as the proportion of patients achieving a best overall response of Complete Response (CR) or Partial Response (PR) according to RECIST criteria
Disease Control Rate (DCR) | Up to 14 days following last dose.
  Defined as the proportion of patients achieving CR, PR, or Stable Disease (SD) as their best overall response.
Duration of Response (DoR) | Up to 14 days following last dose.
  Applicable only to patients with CR or PR, defined as the time from the first documented response to the date of disease progression (PD) or death.
Progression-Free Survival (PFS) | Up to 14 days following last dose.
  The time from the initiation of the first study drug treatment to the occurrence of disease progression or death
Cmax | Single-dose administration on Day 1
  Peak Plasma Concentration (Cmax) of ZX-8177 following a single dose
time to peak concentration (Tmax) | Single-dose administration on Day 1.
  Time to peak concentration (Tmax) of ZX-8177 following a single dose
Area under the concentration-time curve during the dosing interval (AUC0-tau) | Single-dose administration on Day 1.
  Area under the concentration-time curve during the dosing interval (AUC0-tau) of ZX-8177 following a single dose
Trough concentration (Cmin) | Up to 1 hour before the first dose on Cycle 2 Day 1 (each cycle is 28 days).
  Trough concentration (Cmin) of ZX-8177 following multiple doses
Cmax | Up to 1 hour before the first dose on Cycle 2 Day 1 (each cycle is 28 days).
  Peak Plasma concentration (Cmax) of ZX-8177 following multiple doses
Area under the concentration-time curve over the dosing interval (AUC0-tau) | Up to 1 hour before the first dose on Cycle 2 Day 1 (each cycle is 28 days).
  Area under the concentration-time curve over the dosing interval (AUC0-tau) of ZX-8177 following multiple doses
Time to peak concentration (Tmax) | Up to 1 hour before the first dose on Cycle 2 Day 1 (each cycle is 28 days).
  Time to peak concentration (Tmax) of ZX-8177 following multiple doses
accumulation ratio for Cmax (Rac_Cmax) | Up to 1 hour before the first dose on Cycle 2 Day 1 (each cycle is 28 days).
  Accumulation ratio for Cmax (Rac_Cmax) of ZX-8177 following multiple doses
Accumulation ratio for AUC0-tau (Rac_AUC0-tau) | Up to 1 hour before the first dose on Cycle 2 Day 1 (each cycle is 28 days).
  Accumulation ratio for AUC0-tau (Rac_AUC0-tau) of ZX-8177 following multiple doses
Changes in CXCL10 in the blood during the treatment process. | Up to 30 days following last dose.
  Changes in CXCL10 in the blood during the treatment process.
Changes in CXCL9 during the treatment process | Up to 30 days following last dose.
  Changes in CXCL9 during the treatment process
Changes in GZMB during the treatment process | Up to 30 days following last dose.
  Changes in GZMB during the treatment process
Changes in IL6 during the treatment process | Up to 30 days following last dose.
  Changes in IL6 during the treatment process
Changes in MCP-1 during the treatment process | Up to 30 days following last dose.
  Changes in MCP-1 during the treatment process
Changes in TNF during the treatment process | Up to 30 days following last dose.
  Changes in TNF during the treatment process

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai GoBroad Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No